CLINICAL TRIAL: NCT02561065
Title: Long-term Impact Evaluation of a Worksite-based Lifestyle Intervention to Reduce Cardiovascular Risk in Office Workers
Acronym: TANSNIP-PESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Instituto de Salud Carlos III (Other Government); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TANSNIP CNIC-VUMC-SANTANDER
Record Dates: First submitted 2015-05-27; First posted 2015-09-25 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-03

CONDITIONS: Atherosclerosis
Keywords: Health Lifestyle; Lifestyle Risk Reduction; Health Behavior; Sedentary Lifestyle; Intervention Studies; Cardiovascular risk in office workers; Motivational Interview; Preventive health services; Health education; Physical activity; Dietary behaviour intervention; Workplace
MeSH Terms: conditions — Atherosclerosis; Risk Reduction Behavior; Health Behavior; Sedentary Behavior; Health Education; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lifestyle intervention high risk group. (Experimental): Participants in the intervention group will receive the intervention on top of standard care.
  Interventions: Behavioral: Lifestyle intervention
- Standard care high risk group. (No Intervention): Each participant in the standard care group will receive care as usual, provided by his own occupational physician (OP) and other possible care providers.
- Lifestyle intervention low risk group. (Experimental): Participants in the intervention group will receive the intervention on top of standard care.
  Interventions: Behavioral: Lifestyle intervention
- Standard care low risk group. (No Intervention): Each participant in the standard care group will receive care as usual, provided by his own occupational physician (OP) and other possible care providers.

INTERVENTIONS:
Behavioral: Lifestyle intervention — 1. Each participant will receive 12 personalized lifestyle counseling sessions given face-to-face by a trained practitioner.
  2. The Fitbit physical activity tracker gives summaries of the participant's physical activity, provides stimulating prompts and rewards, and allows for social media sharing and competition.
  3. A Sit-stand workstation allows to adjust the height of the participant workstation, including the computer screen, keyboard and mouse and allows them to easily switch between sitting and standing throughout the workday.
  Arms: Lifestyle intervention high risk group.; Lifestyle intervention low risk group.

SUMMARY:
The main objective of TANSNIP-PESA is to determine in a population of asymptomatic bank employees with high and low imaging defined cardiovascular disease (CVD) risk the effectiveness of a comprehensive 3-year worksite-based lifestyle intervention consisting of 12 personalized lifestyle counseling sessions, a Fitbit physical activity tracker and a sit-stand Workstation.

DETAILED DESCRIPTION:
We will study the effectiveness of a 30-month worksite-based lifestyle program aimed to promote cardiovascular health in participants having a high or a low degree of subclinical atherosclerotic plaque burden (SAPB), compared to standard care.

Methods: We will conduct a randomized controlled trial (RCT) including middle-aged bank employees from the ´Progression of Early Subclinical Atherosclerosis´ (PESA) cohort, stratified by SAPB. Within each stratum, participants will be randomized 1:1 to receive a lifestyle program or standard care.

The primary outcome measure is the adapted FUSTER-BEWAT CVD risk and lifestyle composite score and secondary outcome measures include physical activity, sedentary time, standing time, diet, smoking, anthropometric measures, blood biomarkers, self-rated health, work-related outcomes, healthcare consumption, program process measures and cost measures.

ELIGIBILITY:
Inclusion Criteria:

1. Employees aged 40 to 60 years of the PESA (Progression of Early Subclinical Atherosclerosis) cohort study (48) from the Banco de Santander Headquarters in Madrid (Spain).
2. Employees to be included need to be 1 year before PESA 2/3 visit (-1/ +2 months deviation).
3. Employees that can be stratified into a high or low degree of imaging defined SAPB. High degree of imaging-defined SAPB will be defined as a high burden of atherosclerotic disease detected either by 2D ultrasound (upper tertile sum of maximum thickness of the plaques or coronary artery calcium score (CACS) by computed tomography ≥ 1 point). Low degree of imaging-defined SAPB will be defined as having a CACS Agatston score of zero and no plaque by 2D ultrasound or being in the lowest two tertiles of plaque burden. Participants without plaque burden but with a BMI ≥ 25, or; reporting at least one unhealthy lifestyle behavior in their last PESA visit (i.e., <150 min/wk of at least moderate intensity physical activity assessed by accelerometer, sitting >7 h/d as assessed by accelerometer, not meeting Mediterranean diet guidelines as assessed by a computerized dietary history tool previously developed and validated in the EPIC-Spain study and improved by ENRICA investigators, or smoking) will also be included in the low SAPB group.

Exclusion Criteria:

1. Prior history of cardiovascular disease (myocardial infarction, angina pectoris, stroke, peripheral vascular disease, aortic aneurysm, angioplasty, heart surgery, atrial fibrillation, or any other heart disease).
2. Active treatment for cancer, history of transplant with active immunosuppressive or immunomodulator treatment.
3. Morbid obesity (body mass index ≥40 kg/m2).
4. Presence of any disease that decreases life expectancy to 3 years, or any condition that could affect adherence to the study procedures.
5. Participants are also excluded if they are pregnant or lactating women.
6. Employees without plaque burden, a healthy BMI and a healthy lifestyle will be excluded from the RCT.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1020 (Actual)
Dates: Start 2015-05-25 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Adapted FUSTER-BEWAT score (Blood pressure, Physical activity, Sedentary time, Body Mass Index, Fruit and Vegetable Consumption and Smoking). | Changes between baseline, and Year 1, and Year 2 and Year 3.
  Composite score consisting of: Blood pressure, Physical activity, Sedentary time, Body Mass Index, Fruit and Vegetable Consumption (as a proxy for overall diet) and Smoking.

SECONDARY OUTCOMES:
Original FUSTER-BEWAT score. | Changes between baseline, and Year 1, and Year 2 and Year 3.
  The initial FUSTER-BEWAT score will also be calculated in addition as a secondary outcome for future testing of psychometric properties of the adapted FUSTER-BEWAT score
Objective physical activity/sedentary time. | Changes between baseline, and Year 1, and Year 2 and Year 3
  Physical activity and sedentary time will be objectively assessed with an activPAL activity monitor (PAL technologies Limited, Glasgow, UK). Participants will also complete a short daily diary, reporting the exact wearing times.
Self-reported lifestyle behaviors. | Changes between baseline, and Year 1, and Year 2 and Year 3
  The following questionnaires regarding physical activity and sedentary behavior will be administered: the International Physical Activity Questionnaire (IPAQ short form) (also at 4 and 6 months); the Occupational Sitting and Physical Activity Questionnaire (OSPAQ) (also at 4 and 6 months); the Workforce Sitting Questionnaire (WSQ) (also at 4 and 6 months); and single questions to assess average daily standing.
  Data on dietary habits will be collected (also at 4 months) with the Mediterranean Diet Adherence Screener (MEDAS).
  Smoking status will be a self-reported measure, as well as the average number of cigarettes or other tobacco products consumed daily.
  Further, sleeping will be measured using the Sleep Habits Questionnaire developed by the Sleep Heart Health Study.
Physical assessments. | Changes between baseline, and Year 1, and Year 2 and Year 3.
  Waist circumference, body height, body weight, and blood pressure.
Cardio-metabolic biomarkers. | Changes between baseline, and Year 1, and Year 2 and Year 3.
  Complete blood count and chemistry panel as well as specific biomarkers related to subclinical atherosclerosis will be obtained.
Psychosocial assessment. | Changes between baseline, and Year 1, and Year 2 and Year 3.
  Depression will be measured using the Center for Epidemiologic Studies Depression Scale (CES-D). Perceived stress will be measured using the Perceived Stress Scale (PSS).
  Social support will be measured using the official Spanish translated ENRICHD Social Support Instrument (ESSI).
  Job strain will be measured with an adapted version of the official Spanish translation of the Job Content Questionnaire (JCQ).
  Quality of life will be self-reported using the EuroQol (EQ-5D-5L). Relaxation and detachment after work will be measured using the Recovery Experience Questionnaire.
  Self-rated health will be assessed with the EuroQol Visual Analogue Scale (EQ VAS).
  Vitality will be measured using the Vitality questionnaire (VITA-16).
Personal characteristics. | Changes between baseline, and Year 1, and Year 2 and Year 3.
  Sociodemographic information, including age, gender, marital status, working hours per week, employment status, job type, income and education level, will be assessed.
Economic evaluation. | Changes between 4 months up to 36 months (every 3 months measured).
  To evaluate the cost-effectiveness of the lifestyle program, sickness absenteeism, presenteeism (i.e., working while feeling ill) and healthcare consumption (e.g. general practitioner, allied health professionals, complementary medicine consumption) will be assessed every 3 months until 36 months after baseline. Sickness absenteeism and presenteeism will be assessed with items from the WHO Health and Work Performance Questionnaire (WHO-HPQ). Presenteeism is conceptualized in the WHO-HPQ as a measure of actual work performance in relation to best performance, irrespective of the presence or absence of health complaints. Sickness absenteeism will be self-reported using the WHO-HPQ in hours per month.
Intervention process measures. | Changes between baseline, 4 months and Year 1, and Year 2 and Year 3
  Feasibility of the program using quantitative and qualitative methods on three levels: the participant, the psychologist and the stakeholder.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD, PhD, Study Chair — Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III; Jose Maria Castellano, MD, PhD, Principal Investigator — Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III; Hidde van der Ploeg, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Willem van Mechelen, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Borja Ibañez, MD, PhD, Principal Investigator — Centro Nacional de Investigaciones Cardiovasculares Carlos III (F.S.P.); Antonio Fernandez-Ortiz, MD, PhD, Principal Investigator — Centro Nacional de Investigaciones Cardiovasculares Carlos III (F.S.P.); Ines García Lunar, MD, PhD, Principal Investigator — Centro Nacional de Investigaciones Cardiovasculares Carlos III (F.S.P.)

REFERENCES:
- [Derived] Garcia-Lunar I, van der Ploeg HP, Fernandez Alvira JM, van Nassau F, Castellano Vazquez JM, van der Beek AJ, Rossello X, Fernandez-Ortiz A, Coffeng J, van Dongen JM, Mendiguren JM, Ibanez B, van Mechelen W, Fuster V. Effects of a comprehensive lifestyle intervention on cardiovascular health: the TANSNIP-PESA trial. Eur Heart J. 2022 Oct 11;43(38):3732-3745. doi: 10.1093/eurheartj/ehac378. PMID 35869885
- See also: A 30-month worksite-based lifestyle program to promote cardiovascular health in middle-aged bank employees: Design of the TANSNIP-PESA randomized controlled trial — https://www.ncbi.nlm.nih.gov/pubmed/?term=TANSNIP